CLINICAL TRIAL: NCT00459160
Title: A Comparison of Two Target Mean Arterial Pressures in the Resuscitation of Hypotensive Trauma Patients Undergoing Laparotomy or Thoracotomy for Trauma: A Prospective Randomized Controlled Clinical Trial
Brief Title: A Comparison of Two Target Mean Arterial Pressures in the Resuscitation of Hypotensive Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Matthew M. Carrick, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (ER) H-19631
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Hemorrhagic Shock; Trauma; Wounds, Penetrating; Shock, Traumatic; Multiple Trauma
Keywords: Hypotensive Resuscitation; Hypotensive Anesthesia; Hemorrhagic Shock; Penetrating Trauma
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries; Wounds, Penetrating; Shock, Traumatic; Multiple Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low MAP Group (Experimental): Hypotensive Group with a target minimum MAP of 50 mmHg
  Interventions: Procedure: Intraoperative Hypotensive Resuscitation
- High MAP group (No Intervention): Non experimental group: These patients will have a target minimum MAP of 65 mm Hg

INTERVENTIONS:
Procedure: Intraoperative Hypotensive Resuscitation — Patients will have a target minimum MAP of 50 for the case
  Arms: Low MAP Group

SUMMARY:
The goal of this study will be to determine if a lower than normal blood pressure during surgery for bleeding in the abdomen or chest will result in decreased bleeding and decreased chance of death.

DETAILED DESCRIPTION:
For the proposed study, all trauma patients undergoing laparotomy or thoracotomy for trauma that had a systolic blood pressure < 90 mmHg prior to going to the operating room will be randomized to one of two groups. The randomization will take place at the operating room door. The first group will have a target minimum mean arterial pressure of 50 mm Hg (LMAP) and the second group will have a target minimum mean arterial pressure of 65 mmHg (HMAP). Before the operating room and in all other aspects of their care the patients will be treated as per standard of care. Patients will then be followed to determine if there is a difference in 30 day survival between the two groups. Secondary outcome measures will be Sequential Organ Failure Assessment (SOFA) score, APACHE II, ARDS, ICU length of stay, myocardial ischemia, stroke, acidosis, coagulopathy by conventional labs and thromboelastogram, estimated blood loss, transfusion requirements, Glasgow Outcome Score, the presence of leukocyte apoptosis, the serum level of the pro-inflammatory cytokines, IL-6 and G-CSF, and the rate of infectious complications (VAP, UTI, Wound infections). Blood samples (20 ml each) will be taken at three time points: prior to randomization, immediately after the end of resuscitation protocol, and 24 hrs after randomization. Blood will be examined for the presence of leukocyte apoptosis and levels of IL-6 and G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients seen in the Ben Taub emergency center that have suffered a trauma, have a systolic blood pressure less than 90mm Hg, and are going to the operating room for a laparotomy or thoracotomy

Exclusion Criteria:

* Known or suspected head injury
* Age > 45 years old, <= 12 years old
* Incarcerated individuals
* Pregnant women
* Patients with an advanced directive that refuse resuscitation
* Patients with "opt-out" bracelets that signify their refusal of participation in the project

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 271 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
30 day survival | 30 days

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score | 30 days
APACHE II | 30 days
ARDS | 30 days
ICU length of stay | 30 days
Ventilator-free days | 30 days
Myocardial ischemia | 30 days
Stroke | 30 days
Acidosis (pH and BE) | 30 days
Coagulopathy by conventional labs and thromboelastogram | 30 days
Estimated blood loss | 30 days
Transfusion requirements | 30 days
Glasgow Outcome Score | 30 days
Quantification of leukocyte apoptosis | 2 days
Rate of infectious complications (VAP, UTI, wound infections). | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Carrick, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States